CLINICAL TRIAL: NCT02579785
Title: Using mHealth to Promote Post-Menstrual Regulation Contraceptive Uptake and Continuation in the Sylhet, Chittagong and Dhaka Regions of Bangladesh
Brief Title: Using mHealth to Promote Post-Menstrual Regulation Contraceptive Uptake and Continuation in Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marie Stopes International (Other)
Collaborators: Ipas (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MSI-007-14
Record Dates: First submitted 2015-10-16; First posted 2015-10-20 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Contraception; Post-abortion; Abortion
Keywords: Family Planning; Abortion; mHealth; Behaviour Change Communication; Menstrual Regulation; Postabortion; Bangladesh

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- mhealth intervention (Experimental): Receives standard care which includes face to face post-MR family counselling and provision of existing hotline phone number. Also receives Mobile phone based intervention for post-abortion contraceptive uptake.
  Interventions: Behavioral: Mhealth intervention
- Standard Care (No Intervention): Receives standard care which includes face to face post-MR family counselling and provision of existing hotline phone number.

INTERVENTIONS:
Behavioral: Mhealth intervention — A series of ten automated interactive voice messages will be delivered to the participant's mobile phone over a period of 4 months. Messages will be targeted to the method of contraception the participant is using (no-method, condoms, pills, injectable, implant, copper coil). Messages will support uptake of contraception among no-method users. Messages will support existing users to continue their method and to use it correctly and will also encourage participants who are not happy with their method to switch to a different method. All messages will end with five options: Press 1 to repeat the message, press 2 to listen to recorded information about methods of contraception, press 3 to speak to a counsellor, press 4 to tell me you're fine, press 5 to stop receiving these messages.
  Arms: mhealth intervention

SUMMARY:
The purpose of this study is to assess whether a mobile phone intervention can be effectively used to improve post menstrual regulation contraceptive uptake and continuation in Bangladesh.

The study will consist of two phases: Phase I: A formative phase to understand barriers to post-abortion contraceptive uptake and continuation and the content and modality of messages most appropriate for women in the study areas; and Phase II: An RCT will be conducted to test the effectiveness of the mHealth intervention developed during the formative phase on contraceptive use.

DETAILED DESCRIPTION:
The proposed study aims to develop and evaluate a mHealth intervention to promote post-abortion contraceptive uptake and continuation among menstrual regulation clients in the Sylhet, Chittagong and Dhaka regions of Bangladesh.

The aim of the formative phase of the study is to develop an interactive two-way messaging service for post-MR clients. The messaging service will deliver information relating to the women's contraceptive method of choice as well as information about other modern contraceptive methods. This part of the study will focus on determining the modality, content, timing, language and acceptability of messaging services for post menstrual regulation clients.

The aim of the RCT phase is to measure the effect of mHealth on uptake or switching to long-acting reversible contraceptives at the 4 month and 12 month follow ups. The investigators expect mHealth to have a positive effect on uptake and a negative effect on discontinuation rates of contraceptive users.

ELIGIBILITY:
Inclusion Criteria:

* Received menstrual regulation services using Manual Vacuum Aspiration (MVA) or Medical Abortion (MA)
* Have a personal mobile telephone
* Agree to receive messages on mobile about family planning
* Provide informed consent for participation

Exclusion Criteria:

* Received anaesthesia for their MVA procedure
* Intend to become pregnant within the next six months
* Intend to use, or for partner to use, a permanent method of contraception (i.e. sterilisation) within the next six months

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 972 (Actual)
Dates: Start 2015-12-19 (Actual); Primary Completion 2016-07-15 (Actual); Study Completion 2016-07-15 (Actual)

PRIMARY OUTCOMES:
Use of long acting and reversible contraceptive at 4 months | 4 months
  Proportion of subjects that self-report using a long acting and reversible contraceptive (coil or implant)

SECONDARY OUTCOMES:
Use of long acting and reversible contraceptive at 2 weeks and 12 months | 2 weeks and 12 months
  Proportion of subjects that self-report using a long acting and reversible contraceptive (coil or implant)
Use of any modern method at 2 weeks, 4 months and 12 months | 2 weeks, 4 months and 12 months
  The proportion of subjects that self report using any effective modern contraceptive method: Modern contraceptive methods are defined according to the WHO as those associated with <10% 12 month pregnancy rates (WHO, 2011)
Pregnancy | 4 months and 12 months
  Proportion of subjects pregnant that self-report pregnancy at the time of follow-up
Menstrual Regulation | 4 months and 12 months
  Proportion of subjects that self report having had an MR procedure since baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Anderson, PhD, Principal Investigator — Ipas; Sadid Nuremowla, PhD, Principal Investigator — Marie Stopes International
Locations (41):
- Bangladesh (41):
  - Marie Stopes Bangladesh Maternity Clinic,, Chittagong
  - Marie Stopes Clinic Brahman Baria, Chittagong
  - Marie Stopes Clinic Chandpur, Comilla, Chittagong
  - Marie Stopes Clinic Chittagong 1, Chittagong
  - Marie Stopes Clinic Comilla, Chittagong
  - Marie Stopes Clinic Cox's Bazar, Chittagong
  - Marie Stopes Clinic Shitakunda, Chittagong
  - Marie Stopes Femi Maternity Clinic, Chittagong
  - RHSTEP Bandarban Clinic, Chittagong
  - RHSTEP Chittagong Medical College Hospital, Chittagong
  - RHSTEP Clinic Khagrachhari, Chittagong
  - RHSTEP Cox's Bazar Sadar Hospital, Chittagong
  - RHSTEP Rangamati Sadar Hospital, Chittagong
  - Faridpur Maternal and Child Welfare Centre, Dhaka
  - Kishoreganj Maternal and Child Welfare Centre, Dhaka
  - Manikganj Maternal and Child Welfare Centre, Dhaka
  - Mari Stopes Clinic Manikgonj, Dhaka
  - Marie Stopes Bashail Maternity Clinic, Dhaka
  - Marie Stopes Clinic Balurmath, Dhaka
  - Marie Stopes Clinic Gazipur, Dhaka
  - Marie Stopes Clinic Kallyanpur, Dhaka
  - Marie Stopes Clinic Kamrangirchar, Dhaka
  - Marie Stopes Clinic Madaripur, Dhaka
  - Marie Stopes Clinic Mymensingh, Dhaka
  - Marie Stopes Clinic Sherpur, Dhaka
  - Marie Stopes Clinic Tongi, Dhaka
  - Marie Stopes Kadamtali Maternity Clinic, Dhaka
  - Marie Stopes Premium 1 Clinic, Dhaka
  - Marie Stopes Premium 2 Clinic, Dhaka
  - Marie Stopes Referal Clinic, Tangail, Dhaka
  - Mohammapur Fertility Services and Training Centre, Dhaka
  - RHSTEP Dhaka Medical College Hospital, Dhaka
  - RHSTEP Faridpur Medical College Hospital, Dhaka
  - RHSTEP Mymensingh Medical College Hospital, Dhaka
  - RHSTEP Sir Salaimullh Medical College Hospital, Dhaka
  - Rupganj UHC Health Unit, Dhaka
  - Marie Stopes Clinic Chatak, Sylhet
  - Marie Stopes Clinic Moulvi Bazar, Sylhet
  - Marie Stopes Sylhet Maternity Clinic, Sylhet
  - RHSTEP Sylhet OAG Osmani Medical College Hospital, Sylhet
  - Shreemongol UHC Health Unit, Sylhet

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730
- [Derived] Reiss K, Andersen K, Pearson E, Biswas K, Taleb F, Ngo TD, Hossain A, Barnard S, Smith C, Carpenter J, Menzel J, Footman K, Keenan K, Douthwaite M, Reena Y, Mahmood HR, Tabbassum T, Colombini M, Bacchus L, Church K. Unintended Consequences of mHealth Interactive Voice Messages Promoting Contraceptive Use After Menstrual Regulation in Bangladesh: Intimate Partner Violence Results From a Randomized Controlled Trial. Glob Health Sci Pract. 2019 Sep 26;7(3):386-403. doi: 10.9745/GHSP-D-19-00015. Print 2019 Sep. PMID 31558596
- [Derived] Reiss K, Andersen K, Barnard S, Ngo TD, Biswas K, Smith C, Carpenter J, Church K, Nuremowla S, Pearson E. Using automated voice messages linked to telephone counselling to increase post-menstrual regulation contraceptive uptake and continuation in Bangladesh: study protocol for a randomised controlled trial. BMC Public Health. 2017 Oct 3;17(1):769. doi: 10.1186/s12889-017-4703-z. PMID 28974209